CLINICAL TRIAL: NCT05467969
Title: Online Teleteaching and Teleassessment on Clinical Procedural Skills Via Multiscreen Display Layout: A Prospective Observational Cohort Study
Brief Title: Teleteaching on Clinical Procedural Skills
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Theddeus O. H. Prasetyono, Principal Investigator, Chairman of Indonesian Clinical Training and Education Centre, Indonesia University
Other Study IDs: Teleteaching
Record Dates: First submitted 2022-07-04; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Competence; Educational Problems
Keywords: Clinical Competence; Education, Distance; Education, Medical; Motor Skills; Teaching

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traditional teaching: A group of participants learned the skills on site
- Teleteaching: A group of participant who joined the workshop synchronously through the online multiscreen display teleconference platform
  Interventions: Behavioral: Teleteaching of procedural skills through the online multiscreen display teleconference platform

INTERVENTIONS:
Behavioral: Teleteaching of procedural skills through the online multiscreen display teleconference platform — Teleteaching of procedural skills include three different techniques through three different workshops. Each of the workshops was delivered by a respected expert faculty and then accompanied by skills assessment subsequently. Three different group of learners joined the workshops on knotting skills, suturing skills and laparoscopic hand-eye coordination skills respectively.
  Groups: Teleteaching

SUMMARY:
This study aims to develop a model of teleteaching and teleassessment for clinical procedural skills, consisted of teleteaching design making and teleteaching intervention was conducted in September 2020 - February 2021 at a tertiary center Dr. Cipto Mangunkusumo Hospital/ Faculty of Medicine Universitas Indonesia.

DETAILED DESCRIPTION:
Six plastic surgery residents and 12 general practitioners voluntarily participated in 3 different workshops. Three workshops on different procedural skill sets were conducted by including surgical knotting skills, suturing techniques and basic laparoscopic hand-eye coordination skills. A group of participants learned the skills on site, while another group joined the workshop synchronously through the online multiscreen display teleconference platform. The teaching effectiveness was assessed using pre-post written test, OSATS, GRS and self-efficacy. Online skills teleassessment was also compared to the asynchronous assessment based on pre-recorded videos.

ELIGIBILITY:
Inclusion Criteria:

* Medical doctors (General Practitioners or Residents in Plastic Surgery Training) who volunteered to join the workhops

Exclusion Criteria:

* Participants who do not consent to join the workshops

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical doctors (General Practitioners or Residents in Plastic Surgery Training)
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Multiscreen display layouts created from multicamera configurations | 2 months
  A set of configuration of multiscreen display layout was arranged using 3 different cameras to represent 3 different point of views, which accommodated the 1st person view, and two different angles of the 3rd person view
Pre-post written test scores | Through study completion, an average of 6 weeks
  Pre-post written tests consisted of questions based on the teaching materials, used specifically to assess participants' knowledge
Objective Structured Assessment of Technical Skills (OSATS) Score | Through study completion, an average of 6 weeks
  Checklisted-points which assessed each participants' performance while doing each procedural skills, such as
Global Rating Scale (GRS) | Through study completion, an average of 6 weeks
  Consisted of 8 points which assessed each participants' overall performance: professional attitude, timing and movement, correct use of the model, flow, appropriate aseptic techique, overall performance, and final outcome

SECONDARY OUTCOMES:
Self Efficacy Scale | Through study completion, an average of 6 weeks
  Consisted of points in which the participants' rated their condifence and performance after doing the procedures

CONTACTS AND LOCATIONS:
Overall Officials: Theddeus Prasetyono, M.D, Ph.D, Principal Investigator — Indonesian Clinical Training and Education Centre (ICTEC), Faculty of Medicine, Universitas Indonesia
Locations (1):
- Indonesia University, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No